CLINICAL TRIAL: NCT05382598
Title: Early Versus Late Renal Replacement Therapy In Mechanically Ventilated Patients With Acute Kidney Injury
Brief Title: Timing of Renal Replacement Therapy In Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4220
Record Dates: First submitted 2022-04-17; First posted 2022-05-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Timing of RRT in Mechanically Ventilated Patients
Keywords: early and late RRT; AKI; Mechanical ventilation
MeSH Terms: interventions — Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early renal replacement therapy (RRT) group (Active Comparator): In this group of patients, RRT will be initiated if the patient either presents with or develops AKI, while mechanically ventilated, provided that he is in stage 2 according to KDIGO classification.
  RRT will not be delayed till the presence of an urgent indication for the procedure.
  A trial of furosemide stress test will be applied before proceeding towards early RRT after volume optimization.
  Interventions: Procedure: Renal replacement therapy
- Late renal replacement therapy (RRT) group (Active Comparator): This group of patients will receive RRT if they develop any of the following indications:
  * Severe hyperkalemia (> 6.5 mEq/L).
  * Oliguria with failed response to diuretics in the presence of life-threatening pulmonary edema requiring high ventilatory settings i.e. PEEP >10 in addition to FiO2 > 50%.
  * Severe metabolic acidosis (PH <7.15).
  * Uremic pericarditis, encephalopathy or coagulopathy.
  Interventions: Procedure: Renal replacement therapy

INTERVENTIONS:
Procedure: Renal replacement therapy — Renal replacement therapy (RRT) will be initiated in the early group for patients who have stage 2 AKI according to KDIGO classification. The late group will have RRT when they develop any of the absolute indications for RRT

SUMMARY:
This is a randomized controlled study that will be conducted on acute kidney injury (AKI) patients, who are mechanically ventilated, to assess the impact of implementation of early renal replacement therapy (RRT) compared to late RRT on patients outcome.

DETAILED DESCRIPTION:
The study subjects will be randomly divided into two groups (arms).

The first one will be patients who will receive early renal replacement therapy (RRT) according to predefined criteria that will be illustrated later.

The other group of patients will be those who receive late RRT according to the absolute indications of emergency hemodialysis i.e. severe hyperkalemia, life-threatening acidosis, uremic encephalopathy or pericarditis in addition to intractable pulmonary edema.

Appropriate randomization technique will be applied. A computer-based program will be used to perform the randomization procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be on invasive mechanical ventilation.
* Patients in AKI stage 2 , according to KDIGO classification.
* Recruited subjects will include either those who present with AKI on their ICU admission or those who develop AKI during their ICU stay

Exclusion Criteria:

* Those who are known to be in grade 5 CKD according to KDIGO classification. All other grades of CKD from 1 to 4 will be included only if they develop or present with stage 2 AKI on top of their CKD grade
* Those who develop AKI due to obstructive or traumatic causes.
* Patients with septic shock who are on high doses of vasopressors or inotropes (norepinephrine infusion more than 1 mcg/kg/minute, dopamine or dobutamine infusion more than 5 mcg/kg/minute).
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
mortality | 28 days
  ICU mortality
ICU length of stay | through study completion, an average of 1 year
  Duration of ICU stay
Weaning of mechanical ventilation | through study completion, an average of 1 year
  duration of mechanical ventilation

SECONDARY OUTCOMES:
RRT dependency | for more than three months
  Persistent need for renal replacement therapy for at least two sessions per week
Renal functions on discharge from ICU | through study completion, an average of 1 year
  creatinine level on day of discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Elsharkawy, Master, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomas ME, Blaine C, Dawnay A, Devonald MA, Ftouh S, Laing C, Latchem S, Lewington A, Milford DV, Ostermann M. The definition of acute kidney injury and its use in practice. Kidney Int. 2015 Jan;87(1):62-73. doi: 10.1038/ki.2014.328. Epub 2014 Oct 15. PMID 25317932
- [Result] Kellum JA, Lameire N, Aspelin P, Barsoum RS, Burdmann EA, Goldstein SL, et al. Kidney disease: Improving global outcomes (KDIGO) acute kidney injury work group. KDIGO clinical practice guideline for acute kidney injury. Kidney Int Suppl 2012;2:1-138
- [Result] Kidney Disease: Improving Global Outcomes (KDIGO) Blood Pressure Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Blood Pressure in Chronic Kidney Disease. Kidney Int. 2021 Mar;99(3S):S1-S87. doi: 10.1016/j.kint.2020.11.003. No abstract available. PMID 33637192
- [Result] Gaudry S, Hajage D, Benichou N, Chaibi K, Barbar S, Zarbock A, Lumlertgul N, Wald R, Bagshaw SM, Srisawat N, Combes A, Geri G, Jamale T, Dechartres A, Quenot JP, Dreyfuss D. Delayed versus early initiation of renal replacement therapy for severe acute kidney injury: a systematic review and individual patient data meta-analysis of randomised clinical trials. Lancet. 2020 May 9;395(10235):1506-1515. doi: 10.1016/S0140-6736(20)30531-6. Epub 2020 Apr 23. PMID 32334654
- [Result] Wald R, Bagshaw SM. The timing of renal replacement therapy initiation in acute kidney injury: is earlier truly better?*. Crit Care Med. 2014 Aug;42(8):1933-4. doi: 10.1097/CCM.0000000000000432. No abstract available. PMID 25029128
- [Result] Besen BAMP, Romano TG, Mendes PV, Gallo CA, Zampieri FG, Nassar AP Jr, Park M. Early Versus Late Initiation of Renal Replacement Therapy in Critically Ill Patients: Systematic Review and Meta-Analysis. J Intensive Care Med. 2019 Sep;34(9):714-722. doi: 10.1177/0885066617710914. Epub 2017 Jun 1. PMID 28569129
- [Result] Yang XM, Tu GW, Zheng JL, Shen B, Ma GG, Hao GW, Gao J, Luo Z. A comparison of early versus late initiation of renal replacement therapy for acute kidney injury in critically ill patients: an updated systematic review and meta-analysis of randomized controlled trials. BMC Nephrol. 2017 Aug 7;18(1):264. doi: 10.1186/s12882-017-0667-6. PMID 28784106
- [Result] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972
- [Result] Stawicki SP, Braslow BM, Panebianco NL, Kirkpatrick JN, Gracias VH, Hayden GE, Dean AJ. Intensivist use of hand-carried ultrasonography to measure IVC collapsibility in estimating intravascular volume status: correlations with CVP. J Am Coll Surg. 2009 Jul;209(1):55-61. doi: 10.1016/j.jamcollsurg.2009.02.062. Epub 2009 May 1. PMID 19651063
- [Result] Bersten AD, Handy JM. Oh's intensive care manual. 8th ed. Oxford, U.K.: Elsevier; 2018.
- [Result] Fink MP, Vincent JL, Abraham E, Moore FA, Kochanek P. Textbook of critical care. 7th ed. Philadelphia, PA: Elsevier; 2016.
- [Result] Turner N, Lameire N, Goldsmith DJ, Winearls CG, Himmelfarb J, Remuzzi G. Oxford textbook of clinical nephrology. 4th ed. Oxford, United Kingdom: Oxford University Press; 2016.
- [Result] Goldsmith D, Jayawardene S, Ackland P. ABC of kidney disease. 2nd ed. United Kingdom : BMJ Books; 2013.